CLINICAL TRIAL: NCT07110805
Title: Nutrient And Non-Nutrient Intake, Relative Biomarkers And Their Health Impact In Different Target Populations - The NUTRIPOP-BRIDGE Study
Brief Title: Nutrient And Non-Nutrient Intake, Relative Biomarkers and Their Health Effects In Apparently Healthy Participants
Acronym: NUTRI-BRIDGE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Iolanda Cioffi, Dr, University of Milan
Other Study IDs: 110/23
Record Dates: First submitted 2025-07-24; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Participants With/Without Risk Factors for Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
This observational study aims to provide a comprehensive evaluation of dietary habits, physical activity, biomarkers involved in nutrition, metabolic and inflammatory status as well as intestinal permeability in apparently healthy volunteers aged over 18 years working or studying at the University of Milan. Furthermore, the analysis of the gut microbiota composition along with the omics approaches will be crucial for a better comprehension of the relationship between diet and health status in this population. As part of the OnFoods project (Project code PE00000003, Concession Decree No. 1550 of 11 October 2022 adopted by the Italian Ministry of University and Research, CUP D93C22000890001, Project title "ON Foods - Research and innovation network on food and nutrition Sustainability, Safety and Security - Working ON Foods"), the results will be valuable for suggesting targeted dietary and behavioral guidance in the context of public health policies.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy volunteers
* age ≥ 18 years old

Exclusion Criteria:

* Pregnancy or breastfeeding
* not willing to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both workers and students of the University of Milan aged over 18 years old volunteer to participate by responding to calls for study participation (e.g., a flyer or emails).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dietary intake assessment | At baseline and in 1 month
  Two repeated 24h recalls performed at least 3 weeks apart will be used to assess energy, nutrient and non-nutrient intake.

SECONDARY OUTCOMES:
Anthropometry | At baseline
  Anthropometric measures including weight (in kilograms) and height (in meters) will be measured and combined to report body mass index (BMI) in kg/m^2.
Assessment of fat free mass and fat mass | At baseline
  Bio-Impendence Analysis (BIA) was used to assess fat free mass (FFM) in kg and fat mass (FM) in kg.
Bioelectrical phase angle | At baseline
  Bio-Impendence Analysis (BIA) was used to measure phase angle in degree.
MediLite to assess adherence to Mediterranean Diet | At baseline
  The questionnaire consists of 9 items assessing the daily consumption of fruit, vegetables, cereals, meat and meat products, dairy products, alcohol, and olive oil, and the weekly consumption of legumes and fish. Each item provides a score ranging from 0 to 2 points. The final score ranges from 0 (low adherence) to 18 (high adherence to the Mediterranean diet).
MEDAS to assess adherence to Mediterranean Diet | At baseline
  The questionnaire consists of 14 items evaluating the consumption of olive oil for cooking and dressing; daily intake of vegetables, fruits, butter and red meat; weekly intake of wine, legumes, fish, nuts, sweets, pastries or sugar-sweetened beverages; intake of white meat instead of red or processed red meat and the use of "sofrito" sauce. Each item provides a score ranging from 0 to 1 point. The final score ranges from 0 (low adherence) to 14 (high adherence to the Mediterranean diet).
Assessment of physical activity level | At baseline
  The short form of the International Physical Activity Questionnaire (IPAQ) consists of 7 items, exploring the intensity of physical activity based on metabolic equivalent of task (MET) consumption and sedentary behavior.
Assessment of food consumption based on NOVA classification | At baseline
  The NFFQ (NOVA food frequency questionnaire) consists of 94-item grouped in 9 sections headings: (1) fruit and nuts, (2) vegetables and legumes, (3) cereals and tubers, (4) meat and fish, (5) milk, dairy products, and eggs, (6) oils, fats, and seasonings, (7) sweets and sweeteners, (8) beverages and (9) other. Data are reported as g/day and total daily intake for each NOVA category.
Markers of nutritional status | At baseline
  Serum proteins involved in the assessment of nutritional status including albumin in mg/L and transferrin in mg/L as well as serum iron in mg/L will be evaluated through standardized analytical methods.
Fasting glucose and lipid profile | At baseline
  Markers involved in glucose and lipid metabolisms such as fasting glucose in mg/dl, total cholesterol in mg/dl, LDL-cholesterol in mg/dl, HDL-cholesterol in mg/dl and triglycerides in mg/dl will be evaluated in serum through standardized analytical methods.
Liver function | At baseline
  Markers involved in hepatic functions such as aspartate transaminase in U/L, alanine transaminase in U/L and gamma glutamyl transferase in U/L will be evaluated in serum through standardized analytical methods.
Renal function | At baseline
  Markers involved in renal functions including uric acid, azotemia and creatinine in mg/dl will be evaluated in serum through standardized analytical methods.
Vitamins A, E and carotenoids | At baseline
  Plasma vitamin A and vitamin E in µg/mL as well as bioactive compounds such as carotenoids in µg/mL will be evaluated through standardized analytical methods.
Vitamin D | At baseline
  Plasma vitamin D in ng/mL will be evaluated through standardized analytical methods.
Vitamin B12 and folate | At baseline
  Plasma vitamin B12 in ng/mL and folate in ng/mL will be evaluated through standardized analytical methods.
C-reactive protein | At baseline
  C-reactive protein in mg/L will be measured in serum through standardized analytical methods.
Markers of systemic inflammation | At baseline
  Markers involved in the inflammatory status such as TNF-α in pg/mL, IL-6 in pg/mL will be measured in serum through ELISA kits.
Markers of intestinal permeability | At baseline
  Intestinal permeability will be assessed by analyzing serum zonulin in ng/mL and ZO-1 in ng/mL using ELISA kits.
Marker of intestinal permeability | At baseline
  Serum calprotectin in µg/mL and fecal calprotectin in µg/g will be analyzed.
Microbiota composition | At baseline
  Microbiota composition in fecal samples will be evaluated through 16S rRNA sequencing methods.
Proteomic analysis | At baseline
  Proteomic will be performed on serum samples using Somascan.
Metabolomic analysis | At baseline
  Metabolomic will be performed on urine samples by mass spectrometry.
Cellular DNA damage | At baseline
  To assess damage at the cellular DNA level the Comet assay technique will be employed.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Del Bo' Cristian, Principal Investigator — University of Milan; Prof. Riso Patrizia, Principal Investigator — University of Milan; Prof. Martini Daniela, Principal Investigator — University of Milan; Dr. Cioffi Iolanda, Principal Investigator — University of Milan; Dr. Marino Mirko, Principal Investigator — University of Milan
Locations (1):
- Division of Human Nutrition Department of Food, Environmental and Nutritional Sciences - DeFENS Università degli Studi di Milano, Milan, Italy